CLINICAL TRIAL: NCT07299305
Title: Effect of Low Fermentable, Oligo-, di-, Monosaccharides and Polyols (FODMAP) Diet on Improving Symptoms of Patients With Irritable Bowel Syndrome (Randomized Control Trial)
Brief Title: (FODMAP) Diet on Improving Symptoms of Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Irritable bowel syndrome
Record Dates: First submitted 2025-12-08; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2022-11

CONDITIONS: Irritable Bowel Disease
Keywords: IBS, low FODMAP diet, QOL
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens | interventions — Monosaccharides; polyol; Diet

STUDY DESIGN:
Intervention Model Description: A randomized control trial open-label trial .The study included 93patients in intervention group and 90 patients in control group who newly diagnosed with IBS based on Rome IV criteria and subtypes of IBS included constipation-predominant, diarrhea predominant, mixed, and unspecified.
  The sample was collected by a systematic random sample technique. The sample was classified randomly according to intervention type into two groups (108 each group) by block randomization using sealed Envelope website. The participants were classified into 12 blocks (6 block in each group) each block size 18 list length with allocation ratio 1:1, Study was open-label. There was drop out in both intervention and control group, 15 patients were dropped out from intervention group and 21 from control group so the number of participants which completed the study were 93 in intervention group and 90 in control group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): follow low fermentable- oligo-Di- monosaccharides and polyols(FODMPD) diet as intervention program
  Interventions: Dietary Supplement: Low Fermentable, Oligo-, Di-, Monosaccharides and Polyols (FODMAP) Diet
- Control group (No Intervention): control group were patients with irritable bowel syndrome don't follow any intervention program

INTERVENTIONS:
Dietary Supplement: Low Fermentable, Oligo-, Di-, Monosaccharides and Polyols (FODMAP) Diet — The intervention group was subjected to the intervention (health education about LED) . It was conducted through patient-centered educational sessions and follow-up visits in the form of a personal interview and one to one discussion. Participants' phone number was taken for follow-up. Every 2 weeks, the patients were contacted by telephone to resolve any problems related to dietary management. The educational booklet was handled to the patient, it contained all details about how to apply the low FODMAP diet. The message delivered contained information about: Definition of IBS, diagnosis of IBS, red flags of IBS, management of IBS and role and component of low FODMAP diet in IBS. The control group received the educational booklet at the end of the study for ethical purposes.Patients in the intervention group only were asked to fill out the 3 questionnaires related to food acceptability and adherence: FODMAP Adherence Report Scale (FARS), LFD acceptability questionnaire and Food
  Arms: Intervention group

SUMMARY:
Irritable bowel syndrome (IBS) is a common disorder of gut-brain interaction, characterized by chronic abdominal pain and altered bowel habits. A low-FODMAP diet (LFD), which restricts specific types of fermentable carbohydrates, significantly reduces IBS symptoms and improves quality of life (QoL). Objectives: To evaluate the short- and long-term effects of LFD on improving symptom severity and the quality of life of IBS patients attending the family medicine outpatient clinic, and to assess LFD acceptability and adherence of IBS patients. Methods: Randomized control trial conducted on (123 patients) with IBS attending outpatient clinic of family medicine at Tenth of Ramadan University Hospital from 1st of June 2024 to the end of June 2025. An intervention group (No=93) received patient-centered education about LFD, and a control group (No.=90). Participants in both groups underwent an assessment of their BMI, Irritable Bowel Syndrome- Severity Scoring System (IBS-SSS), and irritable bowel syndrome-Quality of Life Measure (IBS-QOL) preintervention during the first visit and reassessed post-intervention after one, three, and six months. Additionally, Patients in the intervention group were assessed for the FODMAP Adherence Report Scale (FARS), LFD acceptability questionnaire, and Food-related QOL questionnaire at one, three-, and six-month post-intervention phases.

DETAILED DESCRIPTION:
A randomized control trial open-label trial was conducted from 1st June 2024 to the end of June 2025 at the family medicine clinic, Tenth of Ramadan University Hospital- Sharkia governorate. It was selected due to the high rate of attendance and the availability of repeated follow-up visits. The study was conducted in accordance with CONSORT guidelines, and a flowchart was used to illustrate the participant selection and allocation process.

The study included 93patients in intervention group and 90 patients in control group who newly diagnosed with IBS based on Rome IV criteria and subtypes of IBS included constipation-predominant, diarrhea predominant, mixed, and unspecified, according to Bertin et al., (2024), aged 18 to 60 years old of both genders, after taking their consent to participate. Exclude Patients who previously diagnosed with GI comorbidities, such as inflammatory bowel disease, celiac disease, lactose malabsorption, significant diverticular disease, or a history of bowel resection, Clinically significant systemic disease, pregnant or lactating, drug abuse, serious psychiatric diseases, or eating disorders, Presence of blood or pus in stool analysis, Individuals with IBS-alarming symptoms as (did not have a normal colonoscopy).

- Sample size: Assuming IBS severity score after 6 weeks was 153+136 vs. 199+102 in LFD VS LGG diet according to (Pedersen et al., 2014), at 80% power and 95 % CI, the estimated sample was 216 cases, 108 cases in each group using the open epi program version 6 at C.I 95%.

- Sampling technique: The sample was collected by a systematic random sample technique. The sample was classified randomly according to intervention type into two groups (108 each group) by block randomaization using sealed Envelope website. The participants were classified into 12 blocks (6 block in each group) each block size 18 list length with allocation ratio 1:1, Study was open-label. There was drop out in both intervention and control group, 15 patients were dropped out from intervention group and 21 from control group so the number of participants which completed the study were 93 in intervention group and 90 in control group.

Study methods:

The study conducted was carried out through 3 phases:

1. st phase (pre intervention) consisted of 3 sections:

   Section I: An inter¬viewing questionnaire was designed to collect data from both group (intervention and control group) include:
   1. Sociodemographic characteristics (Fahmy et al., 2015) .
   2. Assessment Irritable bowel syndrome- severity scoring system (IBS-SSS): The IBS-SSS is a 5-question assessment to appraise the severity, frequency of abdominal pain, intensity of abdominal distention, frustration with bowel habits, and intrusion in quality of life 10 days ago (Francis et al., 1997).
   3. Irritable Bowel Syndrome-Quality of Life Measure (IBS-QOL): The IBS-QOL is a self-report quality-of-life measure specific to IBS that can be used to assess the impact of IBS and its treatment. It consists of 34 items, each with a five-point response scale (Andrae et al., 2013).

   The following questionnaires were used to collect data from intervention group only:

   d. FODMAP Adherence Report Scale (FARS): This evaluates how much the patient adhered to the diet. It consists of 5 questions, each offering five possible answers (always, often, sometimes, rarely, and never) (Maagaard et al., 2016).

   e. LFD acceptability questionnaire: It is composed of 13 items adapted from the nutrition-related QOL (Quality of Life) questionnaire. This investigates the impact of the diet on everyday life. The answers are categorized using 3 possible answers (agree, neutral, and disagree) (Bellini et al., 2020).

   f. Food-related QOL questionnaire: A seven-item questionnaire, based on a 3-point Likert scale, investigating the relationship with food and meals (Bellini et al., 2020) Section II: Stool analysis: to exclude the presence of pus or blood in the stool.

   Section III: Assessment of anthropometric measurements: (Weight, height, and BMI) of the patients Validation of the questionnaires was made as follows: the questionnaires were translated using a back-translation technique. An expert translated the original questionnaires from English into Arabic. The Arabic version of the questionnaires was translated back into English by a bilingual individual. reliability test was done using the reliability coefficients, which was high and suitable for scientific purposes (Cronbach's alpha ranged from 0. 80 to 0.90).
2. nd phase (Intervention phase): The intervention group was subjected to the intervention (health education about LED) versus the control group didn't take intervention. It was conducted through patient-centered educational sessions and follow-up visits in the form of a personal interview and one to one discussion. Participants' phone number was taken for follow-up. Every 2 weeks, the patients were contacted by telephone to resolve any problems related to dietary management. The educational booklet was handled to the patient, it contained all details about how to apply the low FODMAP diet. The message delivered contained information about: Definition of IBS, diagnosis of IBS, red flags of IBS, management of IBS and role and component of low FODMAP diet in IBS. The control group received the educational booklet at the end of the study for ethical purposes.
3. rd phase (Post intervention phase):

After 1st, 3rd, 6th month of the intervention:

Patients in both groups were assessed for their BMI and asked to refill out the same questionnaires in preintervention phase. Patients in the intervention group only were asked to refill out the last 3 questionnaires related to food acceptability and adherence: FODMAP Adherence Report Scale (FARS), LFD acceptability questionnaire and Food-related QOL questionnaire.

Primary outcome: was improvement in IBS severity symptoms score (IBS-SSS), irritable bowel syndrome-Quality of Life Measure (IBS-QOL).

Secondary outcome: was improvement in BMI.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed with IBS based on Rome IV criteria and subtypes of IBS included constipation-predominant, diarrhea predominant, mixed, and unspecified,
* aged 18 to 60 years old of both genders,
* after taking their consent to participate

Exclusion Criteria:

* Patients who previously diagnosed with GI comorbidities (such as inflammatory bowel disease, celiac disease, lactose malabsorption, significant diverticular disease, or a history of bowel resection)
* Clinically significant systemic disease
* pregnant or lactating
* drug abuse
* serious psychiatric diseases
* eating disorders
* Presence of blood or pus in stool analysis
* Individuals with IBS-alarming symptoms as (did not have a normal colonoscopy)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 183 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-10-30 (Actual)

PRIMARY OUTCOMES:
Irritable Bowel Syndrome-Quality of Life Measure (IBS-QOL) | 6 months
  The IBS-QOL is a self-report quality-of-life measure specific to IBS that can be used to assess the impact of IBS and its treatment. It consists of 34 items, each with a five-point response scale ( preintervention, postintervention at 1st, 3rd and 6th month)
IBS severity symptoms score (IBS-SSS) | 6 months
  The IBS-SSS is a 5-question assessment to appraise the severity, frequency of abdominal pain, intensity of abdominal distention, frustration with bowel habits, and intrusion in quality of life 10 days ago ( preintervention and postintervention at 1st month, 3rd month, 6th month

SECONDARY OUTCOMES:
Body Mass Index | 6 months
  Pre and Post measurements of Body mass index(Kg/m^2) at 1st , 3rd, 6th months

CONTACTS AND LOCATIONS:
Overall Officials: Hanaa A Nofal, MD, Study Director — Zagazig University Faculty of Human Medicine
Locations (1):
- Zagazig University outpatients clinics, Zagazig, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: No
Due to privacy of data

REFERENCES:
- [Result] Abdallah, A. M., & Sharafeddin, M. A. Subjective sleep quality among patients with irritable bowel syndrome attending an outpatient clinic in Zagazig University Hospital. Egypt. J. Community Med.2021, 39(1), 23-31. https://doi.org/10. 21608/ ejcm.2021.144069. Nanayakkara, W. S., Skidmore, P. M., O'Brien, L., Wilkinson, T. J., and Gearry, R. B. Efficacy of the low FODMAP diet for treating irritable bowel syndrome: the evidence to date. Clinical and Experimental Gastroenterology.2016. 9, 131. Ng, Q. X., Yaow, C. Y. L., Moo, J. R., Koo, S. W. K., Loo, E. X. L., et al. A systematic review of the association between environmental risk factors and the development of irritable bowel syndrome. J. Gastroenterol. Hepatol.2024. https://doi.org/10. 1111/ jgh.16587. Barbara, G., Cremon, C., Bellini, M., Corsetti, M., Di Nardo, G., et al. Italian guidelines for the management of irritable bowel syndrome: Joint consensus from the Italian societies of gastroenterology and endoscopy (SIGE), neurogastroenterology and motility (SINGEM), hospital gastroenterologists and endoscopists (AIGO), digestive endoscopy (SIED), general medicine (SIMG), gastroenterology, hepatology and pediatric nutrition (SIGENP), and pediatrics (SIP). Dig. Liver Dis.2023, 55, 187-207. https://doi.org/10.1016/j.dld.2022.10.013. Lusetti, F., Schiepatti, A., Scalvini, D., Maimaris, S., & Biagi, F. Efficacy of a Low-FODMAP Diet for Coeliac Patients with Persistent IBS-like Symptoms despite a Gluten-Free Diet: A Systematic Review. Nutrients.2024. 16(7), 1094. https://doi.org/10. 3390/nu16071094. Van Lanen, A. S., de Bree, A., & Greyling, A. Efficacy of a low-FODMAP diet in adult irritable bowel syndrome: a systematic review and meta-analysis. Eur J Nutr.2021. 60, 3505-22. https://doi.org/10. 1007/s00394-020-02473-0. Bertin, L., Zanconato, M., Crepaldi, M., Marasco, G., Cremon, C., et al. The role of the FODMAP diet in IBS. Nutrients.2024. 16(3), 370. https://doi.org/10.3390/nu16030370.